CLINICAL TRIAL: NCT01666002
Title: Treatment of Onychomycosis Using a 0.65 Millisecond Pulsed Nd:YAG 1064 nm Laser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jean Yuh Tang, Assistant Professor of Dermatology, Stanford University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Onycho-2012
Record Dates: First submitted 2012-08-10; First posted 2012-08-16 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 1. st visit: Patient will come into clinic for initial laser treatment with Nd:YAG 1064 nm laser fitted with special handpiece.
  2. nd visit: 2 weeks after initial laser treatment, patient will be seen for second treatment with Nd:YAG 1064 nm laser fitted with special handpiece.
  Interventions: Device: Laser Treatment (Pulsed Nd:YAG 1064 nm Laser)
- Placebo (No Intervention): 1. st visit: For the control group, no treatment will be given.
  2. nd visit: 2 weeks after initial visit, patient will be seen for second visit

INTERVENTIONS:
Device: Laser Treatment (Pulsed Nd:YAG 1064 nm Laser) — 0.65 Millisecond Pulsed Nd:YAG 1064 nm Laser
  Arms: Treatment

SUMMARY:
The investigators would like to test the treatment of onychomycosis using a 0.65 millisecond pulsed 1064 nm laser fitted with a special onychomycosis handpiece. The investigators will compare the success rates of those receiving laser treatments with untreated patients. This study will provide a clinical basis for determining the relative effectiveness of an increasingly utilized treatment method.

DETAILED DESCRIPTION:
Current antifungal treatments have low cure rates and numerous side effects. A new treatment method, pulsed laser, has been purported to have high rates of treatment in a much shorter time frame than other treatments. While the treatment method has become increasingly popular, studies of its efficacy are few. The investigators hope to learn the cure rate of a novel treatment that is being used by more and more patients. This knowledge will be essential to physicians as they consider employing this new technology in their treatment methods.

ELIGIBILITY:
Inclusion Criteria:

* Have Onychomycosis on at least one toe.
* Age 18 or older.
* Consent to research use of their toenail clippings.

Exclusion Criteria:

* Current immunosuppression (cancer, autoimmune disease) or taking immunosuppressive drugs.
* Pregnant female.
* Age 75 or older.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-09; Primary Completion 2013-10 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean Tang, MD, PhD, Principal Investigator — Stanford University; Tyler Hollmig, MD, Study Chair — Stanford University; Michael Henderson, BA, Study Director — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hochman LG. Laser treatment of onychomycosis using a novel 0.65-millisecond pulsed Nd:YAG 1064-nm laser. J Cosmet Laser Ther. 2011 Feb;13(1):2-5. doi: 10.3109/14764172.2011.552616. Epub 2011 Jan 21. PMID 21250792
- [Background] Vural E, Winfield HL, Shingleton AW, Horn TD, Shafirstein G. The effects of laser irradiation on Trichophyton rubrum growth. Lasers Med Sci. 2008 Oct;23(4):349-53. doi: 10.1007/s10103-007-0492-4. Epub 2007 Sep 28. PMID 17902014
- [Background] Landsman AS, Robbins AH. Treatment of mild, moderate, and severe onychomycosis using 870- and 930-nm light exposure: some follow-up observations at 270 days. J Am Podiatr Med Assoc. 2012 Mar-Apr;102(2):169-71. doi: 10.7547/1020169. PMID 22461276
- [Result] Kimura U, Takeuchi K, Kinoshita A, Takamori K, Hiruma M, Suga Y. Treating onychomycoses of the toenail: clinical efficacy of the sub-millisecond 1,064 nm Nd: YAG laser using a 5 mm spot diameter. J Drugs Dermatol. 2012 Apr;11(4):496-504. PMID 22453588

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We enrolled adults (18-75 years) with a clinical diagnosis of onychomycosis from the dermatology clinic at Stanford between July and December 2011. The key inclusion criterion was a diagnosis of onychomycosis by clinical toenail morphology confirmed by positive culture.
Pre-assignment Details: Patients were randomized following simple randomization procedures (computerized random number generator) in a 2:1 ratio into laser or control groups.
Groups:
- Treatment: 1. st visit: Patient will come into clinic for initial laser treatment with Nd:YAG 1064 nm laser fitted with special handpiece.
  2. nd visit: 2 weeks after initial laser treatment, patient will be seen for second treatment with Nd:YAG 1064 nm laser fitted with special handpiece.
  Laser Treatment (Pulsed Nd:YAG 1064 nm Laser): 0.65 Millisecond Pulsed Nd:YAG 1064 nm Laser
  42 patients were assessed and 27 met eligibility criteria of a diagnosis of onychomycosis by clinical toenail morphology confirmed by positive culture.
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 17 | 10
Completed | 12 | 10
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 5 | 0

BASELINE CHARACTERISTICS:
Population: Sample size calculations (STATA 10, Stat Corp, College Station, TX) indicated that we needed to enroll 24 patients at a 2:1 ratio for 80% power to detect a minimal proximal nail plate difference of 2.5 mm in the 2 groups with a 2-sided alpha of 0.05.
Groups:
- Treatment: 1. st visit: Patient will come into clinic for initial laser treatment with Nd:YAG 1064 nm laser fitted with special handpiece.
  2. nd visit: 2 weeks after initial laser treatment, patient will be seen for second treatment with Nd:YAG 1064 nm laser fitted with special handpiece.
  Laser Treatment (Pulsed Nd:YAG 1064 nm Laser): 0.65 Millisecond Pulsed Nd:YAG 1064 nm Laser
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 17 | 10 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (14) | 65 (8) | 59 (13)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 4 | 16
  >=65 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 14 | 8 | 22
Region of Enrollment [Number; unit: participants]
  United States | 17 | 10 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Primary End Point Was the Percentage of Patients With a Negative Mycological Culture.
Time Frame: 1 year
Measure: Number; unit: percentage of participants
Groups:
- Treatment: 1. st visit: Patient will come into clinic for initial laser treatment with Nd:YAG 1064 nm laser fitted with special handpiece.
  2. nd visit: 2 weeks after initial laser treatment, patient will be seen for second treatment with Nd:YAG 1064 nm laser fitted with special handpiece.
  Laser Treatment (Pulsed Nd:YAG 1064 nm Laser): 0.65 Millisecond Pulsed Nd:YAG 1064 nm Laser
  After 3 months, 4 of 12 patients (33%) in the laser group had negative fungal cultures. Of the 4 patients in the laser group with baseline cultures positive for a non-dermatophyte mold, 2 (50%) had negative fungal cultures. After 3 months of observation, 2 of 10 (20%) control subjects had negative cultures. Of the 3 patients in the control group with baseline cultures positive for a non-dermatophyte mold, 1 (33%) had a negative fungal culture. There was no significant difference in the percentage of patients with negative nail cultures between laser versus control groups (P = .49).
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 12 | 10
percentage of participants | 12 | 10
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p < 0.05, Chi-squared

2. Secondary Outcome: Proximal Clearance of Fungus on Nail
Description: The secondary end point was proximal nail plate clearance as assessed directly by a single study physician, who measured the clinical involvement defined as total length of abnormal nail per each nail of each of the patients' toenails, and confirmed by digital analysis of toenail photographs with ImageJ software.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: nails
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 10 | 6
Number analyzed (nails) | 39 | 39
mm | 0.44 (1.1) | 0.15 (0.7)
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Groups:
- Treatment: 1. st visit: Patient will come into clinic for initial laser treatment with Nd:YAG 1064 nm laser fitted with special handpiece.
  2. nd visit: 2 weeks after initial laser treatment, patient will be seen for second treatment with Nd:YAG 1064 nm laser fitted with special handpiece.
  Laser Treatment (Pulsed Nd:YAG 1064 nm Laser): 0.65 Millisecond Pulsed Nd:YAG 1064 nm Laser
  No patients reported complications or adverse events after 2 sessions.
Arm/Group | Treatment | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/10
Other Adverse Events (participants affected / at risk) | 0/17 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No